CLINICAL TRIAL: NCT02188095
Title: Post Market Clinical Follow-Up Study of Excia T® Hip Prosthesis
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1401
Record Dates: First submitted 2014-06-26; First posted 2014-07-11 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Hip Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Excia T®

SUMMARY:
Clinical and radiological 10 year results of Excia T® Hip Stem

ELIGIBILITY:
Inclusion Criteria:

* Patient gave written informed consent
* age ≥ 18 years

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2015-10-06 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of the Implant | 10 years
  Kaplan-Meier Survival Rate up to 10 years

SECONDARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score (HOOS) | preoperatively, intraoperatively + discharge, after 3 and 12 months 3, 5 and 10 years
  Documentation of clinical outcome with HOOS Score
Change of functional outcome over follow-up period (Harris Hip Score (HHS)) | at discharge, after 3 and 12 months 3, 5 and 10 years
  The Harris Hip Score (HHS) is one of the most used scores in total hip arthroplasty, mainly combining range of motion questions with questions regarding daily life activities.
Pain Assessment | at 6 examinations during follow-up (discharge, after 3 and 12 months and 3, 5, and 10 years)
  Pain will be measured with a Visual Analogue Scale (VAS), at rest and when walking on flat ground. The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patients are asked to mark their current pain level on the line.
Shaftposition ap and lateral | 10 years
  Radiological documentation of shaftposition in ap and lateral view discharge, after 3 and 12 months and 3, 5, and 10 years
Stress Shielding | 10 years
  Radiological documentation of stress shielding after 3 and 12 months and 3, 5, and 10 years
Hypertrophies | 10 years
  Radiological documentation of hypertrophies after 3 and 12 months and 3, 5, and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aldinger, Prof. Dr., Principal Investigator — Diakonie-Klinikum Stuttgart
Locations (2):
- Germany (2):
  - Vulpius Klinik, Bad Rappenau
  - Diakonie Klinikum Stuttgart, Stuttgart